CLINICAL TRIAL: NCT01047124
Title: Randomised Control Trial of the Clinical and Cost Effectiveness of a Specialist Expert Mood Disorder Team for Refractory Unipolar Depressive Disorder
Brief Title: Trial of the Clinical and Cost Effectiveness of a Specialist Expert Mood Disorder Team for Refractory Unipolar Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09044
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Unipolar Depressive Disorder
Keywords: Depression; Collaborative Care; Cognitive Behaviour Therapy; Mental Health Services; Antidepressants
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Specialist mood disorders team: treatment plan according to need
  Interventions: Other: Specialist Mood Disorders Team
- Treatment as usual (No Intervention)

INTERVENTIONS:
Other: Specialist Mood Disorders Team — The specialist mood disorders team will include a psychiatrist and health professionals providing cognitive behaviour therapy. Together the team will assess participants and then provide a co-ordinated and supervised combination of pharmacological and psychological treatment according to guidelines developed by NICE and the British Association of Psychopharmacology. Each participant will receive a treatment plan that is tailored to his/her specific needs.
  Other Names: Collaborative care for depression
  Arms: Intervention

SUMMARY:
The purpose of this study is determine whether a specialised mood disorder service, which offers tailored psychological and pharmacological treatment, is more effective in the treatment of chronic unipolar depressive disorder then treatment as usual.

DETAILED DESCRIPTION:
A pragmatic randomised controlled trial of a specialist mood disorder intervention versus treatment as usual will be conducted. Patients will be individually randomised with stratification by mental health trust to either treatment by a specialist team offering tailored psychological and pharmacological treatment or treatment as usual.

The specialist mood disorders team will include a psychiatrist and health professionals providing cognitive behaviour therapy. Together the team will assess participants and then provide a co-ordinated and supervised combination of pharmacological and psychological treatment according to guidelines developed by NICE and the British Association of Psychopharmacology. Each participant will receive a treatment plan that is tailored to his/her specific needs. The participants in the treatment as usual team will have their usual access to the same treatments. The outcome in terms of improvement in depressive symptoms, function and costs will be examined after one year in service users with chronic depression.

Eligible patients will be followed for 12 months and the primary outcomes will be observer rated depressive symptoms and cost effectiveness from a health and social care perspective. Along side the RCT, implementation analysis and audit of the standard care and specialised care for depression will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* The responsible medical officer or care coordinator leading care considers the patient to be suffering from a primary unipolar depressive disorder which is not a consequence of having another axis 1 or 2 psychiatric disorder.
* Age over 18 years.
* Able and willing to give oral and written informed consent to participation in the study.
* From the date of first assessment by a health professional working for the index mental health trust, they have been offered or received direct care from one or more health professionals from the Trust three or more occasions for 6 months.
* Meet NICE criteria for moderate depression, namely the presence of five out of nine symptoms of (NICE, 2004), have a Hamilton Depression Rating Scale of at least 20, and score 60 or less on the Global Assessment of Functioning Scale (American Psychiatric Association, 1994).

Exclusion Criteria:

* Is receiving emergency care for suicide risk, risk of severe neglect or homicide risk and requires it; however, patients will not be excluded because of such risk provided the risk is adequately contained with their current care setting and the primary medical responsibility for care remains with the referring team.
* Does not speak fluent English.
* Is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2009-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale - Grid version | 6 months

SECONDARY OUTCOMES:
Change in self rated depression measures: Beck Depression Inventory version 1; Personal Health Questionnaire; Quick Inventory of Depressive Symptomology | 3 months
Cost utility or cost effectiveness using the Euroqol 5D as a measure of quality of life and costs from health and social care and society perspectives. | 6 months
Change in social adjustment (Cooper, Osborn, Gath & Feggetter, 1982), an assessment of social and occupational functioning. | 6 months
Patient satisfaction and patient/doctor relationship | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Morriss, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Derbyshire Mental Health NHS Trust, Derby, Derbyshire
  - Lincolnshire Partnership Trust, Lincoln, Lincolnshire
  - Nottinghamshire Healthcare NHS Trust, Nottingham, Nottinghamshire

REFERENCES:
- [Background] Anderson IM, Ferrier IN, Baldwin RC, Cowen PJ, Howard L, Lewis G, Matthews K, McAllister-Williams RH, Peveler RC, Scott J, Tylee A. Evidence-based guidelines for treating depressive disorders with antidepressants: a revision of the 2000 British Association for Psychopharmacology guidelines. J Psychopharmacol. 2008 Jun;22(4):343-96. doi: 10.1177/0269881107088441. Epub 2008 Apr 15. PMID 18413657
- [Background] Baker R, Reddish S, Robertson N, Hearnshaw H, Jones B. Randomised controlled trial of tailored strategies to implement guidelines for the management of patients with depression in general practice. Br J Gen Pract. 2001 Sep;51(470):737-41. PMID 11593835
- [Background] Gilbody S, Bower P, Fletcher J, Richards D, Sutton AJ. Collaborative care for depression: a cumulative meta-analysis and review of longer-term outcomes. Arch Intern Med. 2006 Nov 27;166(21):2314-21. doi: 10.1001/archinte.166.21.2314. PMID 17130383
- [Background] Greden JF. The burden of disease for treatment-resistant depression. J Clin Psychiatry. 2001;62 Suppl 16:26-31. PMID 11480881
- [Background] Parker GB, Malhi GS, Crawford JG, Thase ME. Identifying "paradigm failures" contributing to treatment-resistant depression. J Affect Disord. 2005 Aug;87(2-3):185-91. doi: 10.1016/j.jad.2005.02.015. PMID 15979725
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Warden D, Rush AJ, Trivedi MH, Fava M, Wisniewski SR. The STAR*D Project results: a comprehensive review of findings. Curr Psychiatry Rep. 2007 Dec;9(6):449-59. doi: 10.1007/s11920-007-0061-3. PMID 18221624
- [Background] Sartorius N. The economic and social burden of depression. J Clin Psychiatry. 2001;62 Suppl 15:8-11. PMID 11444765
- [Background] Schramm E, Schneider D, Zobel I, van Calker D, Dykierek P, Kech S, Harter M, Berger M. Efficacy of Interpersonal Psychotherapy plus pharmacotherapy in chronically depressed inpatients. J Affect Disord. 2008 Jul;109(1-2):65-73. doi: 10.1016/j.jad.2007.10.013. Epub 2007 Dec 11. PMID 18067973
- [Background] Sheldon TA, Cullum N, Dawson D, Lankshear A, Lowson K, Watt I, West P, Wright D, Wright J. What's the evidence that NICE guidance has been implemented? Results from a national evaluation using time series analysis, audit of patients' notes, and interviews. BMJ. 2004 Oct 30;329(7473):999. doi: 10.1136/bmj.329.7473.999. PMID 15514342
- [Derived] Nixon N, Guo B, Kaylor-Hughes C, Simpson S, Garland A, Dalgleish T, Morriss R. Specialist treatment for persistent depression in secondary care: Sustained effects from a multicentre UK study at 24 and 36 months. J Affect Disord. 2024 Jan 15;345:70-77. doi: 10.1016/j.jad.2023.10.105. Epub 2023 Oct 19. PMID 37863366
- [Derived] Thomson L, Barker M, Kaylor-Hughes C, Garland A, Ramana R, Morriss R, Hammond E, Hopkins G, Simpson S. How is a specialist depression service effective for persistent moderate to severe depressive disorder?: a qualitative study of service user experience. BMC Psychiatry. 2018 Jun 15;18(1):194. doi: 10.1186/s12888-018-1708-9. PMID 29902995
- [Derived] Morriss R, Garland A, Nixon N, Guo B, James M, Kaylor-Hughes C, Moore R, Ramana R, Sampson C, Sweeney T, Dalgleish T; NIHR CLAHRC Specialist Mood Disorder Study Group. Efficacy and cost-effectiveness of a specialist depression service versus usual specialist mental health care to manage persistent depression: a randomised controlled trial. Lancet Psychiatry. 2016 Sep;3(9):821-31. doi: 10.1016/S2215-0366(16)30143-2. Epub 2016 Aug 3. PMID 27498098
- [Derived] Morriss R, Marttunnen S, Garland A, Nixon N, McDonald R, Sweeney T, Flambert H, Fox R, Kaylor-Hughes C, James M, Yang M. Randomised controlled trial of the clinical and cost effectiveness of a specialist team for managing refractory unipolar depressive disorder. BMC Psychiatry. 2010 Nov 29;10:100. doi: 10.1186/1471-244X-10-100. PMID 21114826